CLINICAL TRIAL: NCT02392624
Title: XTEND-CIU (Xolair Treatment Efficacy of Longer Duration in Chronic Idiopathic Urticaria): A Phase IV, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Omalizumab Through 48 Weeks in Patients With Chronic Idiopathic Urticaria
Brief Title: A Study of the Efficacy and Safety of Omalizumab Through 48 Weeks in Participants With Chronic Idiopathic Urticaria
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ML29510
Record Dates: First submitted 2015-03-13; First posted 2015-03-19 (Estimated); Results first posted 2018-03-26 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Urticaria
MeSH Terms: conditions — Urticaria | interventions — Omalizumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Omalizumab (Experimental): Participants will receive open-label omalizumab treatment at 300 mg SC Q4W for 24 weeks. After 24 weeks open-label treatment, eligible participants will be randomized to receive omalizumab treatment at 300 mg SC Q4W for next 24 weeks (up to Week 48). Participants randomized to omalizumab may, at the discretion of the investigator, be transitioned from blinded study drug to open-label omalizumab at 300 mg SC Q4W if they experience clinically significant worsening in their CIU (as judged by the investigator). Participants who are transitioned to open-label omalizumab will continue to receive open-label omalizumab as study drug until Week 48.
  Interventions: Drug: Omalizumab
- Placebo (Placebo Comparator): Participants will receive open-label omalizumab treatment at 300 mg SC Q4W for 24 weeks. After 24 weeks open-label treatment, eligible participants will be randomized to receive placebo SC Q4W for next 24 weeks (up to Week 48). Participants randomized to placebo may, at the discretion of the investigator, be transitioned from blinded study drug to open-label omalizumab at 300 mg SC Q4W if they experience clinically significant worsening in their CIU (as judged by the investigator). Participants who are transitioned to open-label omalizumab will continue to receive open-label omalizumab as study drug until Week 48.
  Interventions: Drug: Omalizumab; Drug: Placebo

INTERVENTIONS:
Drug: Omalizumab — Omalizumab 300 mg administered SC Q4W.
  Other Names: Xolair; RO5489789
Drug: Placebo — Placebo matched to omalizumab administered SC Q4W.
  Arms: Placebo

SUMMARY:
This multicenter, randomized, double-blind, placebo-controlled study will evaluate the efficacy and safety of subcutaneous (SC) omalizumab (Xolair) as an add-on therapy through 48 weeks for treatment of H1 antihistamine refractory chronic idiopathic urticaria (CIU). After completing an initial 24-week open-label treatment period with omalizumab 300 milligrams (mg) every 4 weeks (Q4W), participants responding to omalizumab will be randomized at a 3:2 ratio (omalizumab:placebo) to either continue omalizumab or be transitioned to placebo for a further 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CIU refractory to H1 antihistamines at baseline
* Presence of itch and hives for at least 8 consecutive weeks at any time prior to enrollment despite current use of H1 antihistamine treatment (up to four times the approved dose) during this time period
* UAS7 score (range 0-42) ≥ 16 and itch component of UAS7 (range 0-21) ≥ 8 during 7 days prior to baseline
* Participants must have been on a non-sedating H1 antihistamine treatment (up to four times the approved dose) for CIU for at least 3 consecutive days immediately prior to screening visit with continued current use on the day of the initial screening visit
* CIU diagnosis for ≥ 6 months
* Willing and able to complete a daily symptom eDiary for the duration of the study

Exclusion Criteria:

* Treatment with an investigational agent within 30 days of the initial screening visit
* Body weight less than 20 kilograms
* Clearly defined underlying etiology for chronic urticarias other than CIU
* Evidence of a parasitic infection
* Atopic dermatitis, bullous pemphigoid, dermatitis herpetiformis, senile pruritus or other skin disease associated with itch
* Previous treatment with omalizumab within 1 year prior to the initial screening visit
* Participants may not have taken during treatment period or have been taking within 30 days before the initial screening visit any of the following medications or treatments:

regular (daily/every other day during 5 or more consecutive days) systemic corticosteroids, hydroxychloroquine, methotrexate, mycophenolate, cyclosporine, cyclophosphamide, intravenous immunoglobulin G or plasmapheresis

* Regular (daily/every other day) oral doxepin use within 14 days prior to the initial screening visit
* Pregnant or lactating women, or women intending to become pregnant during the study

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2015-05-18 (Actual); Primary Completion 2017-03-09 (Actual); Study Completion 2017-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (40):
- United States (40):
  - Allergy and Asthma Relief Experts, Granada Hills, California
  - Allergy & Asthma Care Center of Southern California, Long Beach, California
  - Dermatology Research Associate, Los Angeles, California
  - Southern California Research Center, Mission Viejo, California
  - Choc Psf, Amc, Orange, California
  - Allergy & Asthma Consultants, Redwood City, California
  - Allergy and Asthma Clinical Research, Inc., Walnut Creek, California
  - IMMUNOe Research Centers, Centennial, Colorado
  - Colorado Allergy & Asthma Centers, Pc, Denver, Colorado
  - Florida Center for Allergy and Asthma Research, Aventura, Florida
  - Florida Ctr-Allergy & Asthma, Miami, Florida
  - Sarasota Clinical Research, Sarasota, Florida
  - University of South Florida, Tampa, Florida
  - Clinical Research Center of Southern Illinois LLC, Shiloh, Illinois
  - Deaconess Clinic, Evansville, Indiana
  - Dawes Fretzin Clinical Res LLC, Indianapolis, Indiana
  - Abraham Research PLLC, Fort Mitchell, Kentucky
  - Dermatology Specialists Research, LLC, Louisville, Kentucky
  - Allergy & Asthma Specialists, PSC, Owensboro, Kentucky
  - Asthma, Allergy & Sinus Center, Baltimore, Maryland
  - Institute for Asthma & Allergy, Chevy Chase, Maryland
  - Respiratory Medicine Research; Institue of Michigan P.L.C., Ypsilanti, Michigan
  - James Q. Del Rosso, DO, LLC, Las Vegas, Nevada
  - Ocean Allergy & Resp Res Ctr, Brick, New Jersey
  - Winthrop University Hospital, Mineola, New York
  - Aair Research Center, Rochester, New York
  - University of Rochester Medical Center; University Dermatology Associates, Rochester, New York
  - Montefiore Medical Group;Department of Medicine, The Bronx, New York
  - Allergy Partners of Western NC, Asheville, North Carolina
  - Allergy & Respiratory Center, Canton, Ohio
  - Bernstein Clinical Research Center Llc, Cincinnati, Ohio
  - Toledo Inst of Clin Research, Toledo, Ohio
  - Vital Prospects Clin Res Pc, Tulsa, Oklahoma
  - Asthma, Nasal Disease, and Allergy Research Center of New England, East Providence, Rhode Island
  - National Allergy and Asthma Research, Charleston, South Carolina
  - Live Oak Allergy & Asthma Clinic, Live Oak, Texas
  - Allergy & Asthma Research Center, San Antonio, Texas
  - Timber Lane Allergy-Asth Res, South Burlington, Vermont
  - O & O Alpan, LLC, Fairfax, Virginia
  - Premier Clinical Research, Spokane, Washington

REFERENCES:
- [Derived] Casale TB, Murphy TR, Holden M, Rajput Y, Yoo B, Bernstein JA. Impact of omalizumab on patient-reported outcomes in chronic idiopathic urticaria: Results from a randomized study (XTEND-CIU). J Allergy Clin Immunol Pract. 2019 Sep-Oct;7(7):2487-2490.e1. doi: 10.1016/j.jaip.2019.04.020. Epub 2019 Apr 26. No abstract available. PMID 31034999

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 206 participants were enrolled in the study, but only 205 participants received at least one dose of any study treatment. Results include only the treated 205 participants.
Groups:
- Omalizumab (Non-Randomized Participants): Participants received open-label omalizumab treatment at a dose of 300 milligrams (mg) via subcutaneous (SC) injection every 4 weeks (Q4W) for 24 weeks. After Week 24, participants did not receive any treatment and only returned for a final follow-up visit (12 weeks after Week 24 visit).
- Omalizumab (Randomized Participants): Participants received open-label omalizumab treatment at a dose of 300 mg via SC injection Q4W for 24 weeks. After 24 weeks of open-label treatment, participants received randomized treatment with omalizumab 300 mg via SC injection Q4W for a further 24 weeks (up to Week 48). Participants, at the discretion of the investigator, could have been transitioned from blinded study drug to open-label omalizumab at a dose of 300 mg via SC injection Q4W if they experienced clinically significant worsening in their chronic idiopathic urticaria (CIU) (as judged by the investigator). Participants who were transitioned to open-label omalizumab continued to receive open-label omalizumab until Week 48.
- Placebo (Randomized Participants): Participants received open-label omalizumab treatment at a dose of 300 mg via SC injection Q4W for 24 weeks. After 24 weeks of open-label treatment, participants received randomized treatment with placebo matching to omalizumab via SC injection Q4W for a further 24 weeks (up to Week 48). Participants, at the discretion of the investigator, could have been transitioned from blinded study drug to open-label omalizumab at a dose of 300 mg via SC injection Q4W if they experienced clinically significant worsening in their CIU (as judged by the investigator). Participants who were transitioned to open-label omalizumab continued to receive open-label omalizumab until Week 48.
Period: Overall Study
Arm/Group | Omalizumab (Non-Randomized Participants) | Omalizumab (Randomized Participants) | Placebo (Randomized Participants)
Started | 71 | 81 | 53
Completed | 0 | 66 | 40
Not Completed | 71 | 15 | 13
Not completed — Withdrawal by Subject | 15 | 12 | 9
Not completed — Adverse Event | 4 | 1 | 2
Not completed — Pregnancy | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Sponsor/Investigator Decision | 2 | 1 | 0
Not completed — Other | 49 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety evaluable population included all participants who received at least one dose of study medication.
Groups:
- Omalizumab (Non-Randomized Participants): Participants received open-label omalizumab treatment at a dose of 300 mg via SC injection Q4W for 24 weeks. After Week 24, participants did not receive any treatment and only returned for a final follow-up visit (12 weeks after Week 24 visit).
- Omalizumab (Randomized Participants): Participants received open-label omalizumab treatment at a dose of 300 mg via SC injection Q4W for 24 weeks. After 24 weeks of open-label treatment, participants received randomized treatment with omalizumab 300 mg via SC injection Q4W for a further 24 weeks (up to Week 48). Participants, at the discretion of the investigator, could have been transitioned from blinded study drug to open-label omalizumab at a dose of 300 mg via SC injection Q4W if they experienced clinically significant worsening in their CIU (as judged by the investigator). Participants who were transitioned to open-label omalizumab continued to receive open-label omalizumab until Week 48.
- Total: Total of all reporting groups
Arm/Group | Omalizumab (Non-Randomized Participants) | Omalizumab (Randomized Participants) | Placebo (Randomized Participants) | Total
Number analyzed (Participants) | 71 | 81 | 53 | 205
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.5 (14.76) | 43.1 (14.68) | 48.5 (13.22) | 44.6 (14.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 60 | 40 | 153
  Male | 18 | 21 | 13 | 52
Race/Ethnicity, Customized [Number; unit: participants]
  Race: American Indian or Alaska Native | 0 | 2 | 0 | 2
  Race: Asian | 0 | 2 | 3 | 5
  Race: Black or African American | 10 | 6 | 7 | 23
  Race: White | 58 | 68 | 42 | 168
  Race: Mixed/Unknown | 3 | 3 | 1 | 7
  Ethnicity: Hispanic or Latino | 20 | 18 | 5 | 43
  Ethnicity: Not Hispanic or Latino | 50 | 63 | 48 | 161
  Ethnicity: Unknown | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced Clinical Worsening in CIU as Assessed by Urticaria Activity Score Over 7 Days (UAS7) (Clinical Worsening: UAS7 Greater Than or Equal to [>/=] 12, Maintained for At Least 2 Consecutive Weeks)
Description: Urticaria activity score (UAS) is a composite diary-recorded score with numeric severity ratings (0=none to 3=intense) for the number of wheals (hives) per 24 hours and the intensity of the pruritus (itch). The total UAS score (sum of the wheal and pruritus scores) ranges from 0 to 6. Due to variations in chronic urticaria disease intensity, assessment of disease activity was based on a weekly (7 days) UAS score called UAS7, that is, the sum of the daily average UASs (average of morning and evening scores), ranging from 0 to 42 per week. A higher score indicates worse disease. Clinical worsening in CIU was defined as UAS7 >/=12 for at least 2 consecutive weeks post-randomization between Weeks 24 and 48.
Time Frame: From randomization (Week 24) to Week 48
Population: Modified Intent-to-Treat (mITT) population included all randomized participants who received at least one dose of blinded study drug, and achieved one post-baseline efficacy assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Omalizumab (Randomized Participants) | Placebo (Randomized Participants)
Number analyzed (Participants) | 81 | 53
percentage of participants | 21.0 [12.7 to 31.5] | 60.4 [46.0 to 73.5]
Statistical Analysis 1: Comparison: Omalizumab (Randomized Participants) vs Placebo (Randomized Participants); For participants who transitioned to open-label omalizumab, data prior to the date of transitioning was used for analysis; Test type: Superiority; p < 0.0001, Chi-squared; Clinical Worsening Rate Difference = -39.4, 95% CI 2-sided [-54.5 to -22.5]

2. Secondary Outcome: Time to Clinical Worsening in CIU as Assessed by UAS7 (Clinical Worsening: UAS7 >/=12, Maintained for At Least 2 Consecutive Weeks)
Description: The UAS is a composite diary-recorded score with numeric severity ratings (0=none to 3=intense) for the number of wheals per 24 hours and the intensity of the pruritus. The total UAS score ranges from 0 to 6. UAS7 is the sum of the daily average UASs (average of morning and evening scores), ranging from 0 to 42 per week. A higher score indicates worse disease. Time to clinical worsening in CIU was defined as the number of weeks from the first double-blind treatment to the first two-week interval with UAS7 >/=12 for both weeks. If clinical worsening did not occur, time to clinical worsening was censored at the end of the last week for which the UAS7 score was not missing and less than (<) 12, prior to last randomized dose + 4 weeks, or the first open-label transition dose, whichever was earlier. Median time to clinical worsening was estimated using Kaplan-Meier analysis and corresponding 95% confidence interval (CI) was computed using the method of Brookmeyer and Crowley.
Time Frame: From randomization (Week 24) to Week 48
Population: Analysis was performed on mITT population.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Omalizumab (Randomized Participants) | Placebo (Randomized Participants)
Number analyzed (Participants) | 81 | 53
weeks | NA [NA to NA] — Median and corresponding 95% CI could not be estimated due to higher number of censored participants. | 12.0 [9.0 to NA] — Upper limit of 95% CI could not be estimated due to higher number of censored participants.
Statistical Analysis 1: Comparison: Omalizumab (Randomized Participants) vs Placebo (Randomized Participants); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Log Rank

3. Secondary Outcome: Percentage of Participants Who Experienced Clinical Worsening in CIU as Assessed by UAS7 (Clinical Worsening: UAS7 Greater Than [>] 6, Maintained for At Least 2 Consecutive Weeks)
Description: The UAS is a composite diary-recorded score with numeric severity ratings (0=none to 3=intense) for the number of wheals per 24 hours and the intensity of the pruritus. The total UAS score ranges from 0 to 6. UAS7 is the sum of the daily average UASs (average of morning and evening scores), ranging from 0 to 42 per week. A higher score indicates worse disease. Clinical worsening in CIU was defined as UAS7 >6 for at least 2 consecutive weeks post-randomization between weeks 24 and 48.
Time Frame: From randomization (Week 24) to Week 48
Population: Analysis was performed on mITT population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Omalizumab (Randomized Participants) | Placebo (Randomized Participants)
Number analyzed (Participants) | 81 | 53
percentage of participants | 32.1 [22.2 to 43.4] | 64.2 [49.8 to 76.9]
Statistical Analysis 1: Comparison: Omalizumab (Randomized Participants) vs Placebo (Randomized Participants); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0004, Chi-squared; Clinical Worsening Rate Difference = -32.1, 95% CI 2-sided [-47.9 to -14.9]

4. Secondary Outcome: Change From Randomization (Week 24) to Week 48 in UAS7 Among Participants Who Received Total 48 Weeks Treatment With Omalizumab
Description: The UAS is a composite diary-recorded score with numeric severity ratings (0=none to 3=intense) for the number of wheals per 24 hours and the intensity of the pruritus. The total UAS score ranges from 0 to 6. UAS7 is the sum of the daily average UASs (average of morning and evening scores), ranging from 0 to 42 per week. A higher score indicates worse disease. A negative change in score (Week 48 score minus Week 24 score) indicates improvement.
Time Frame: Week 24 (randomization) and Week 48
Population: Analysis was performed on participants in mITT population who received total 48 weeks of treatment with omalizumab. If UAS7 data was missing, last observation carry forward (LOCF) method was used post-Week 24 for the closest non-missing UAS7 data up to Week 48.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Omalizumab (Randomized Participants)
Number analyzed (Participants) | 72
units on a scale
  Week 24 (Randomization) | 0.69 (1.448)
  Change at Week 48 | 1.77 (6.470)
Statistical Analysis 1: Comparison: Omalizumab (Randomized Participants); The null hypothesis for this test was that the mean change from Week 24 to Week 48 in UAS7 score was >/=5 and the alternative hypothesis was that the mean change from Week 24 to Week 48 in UAS7 score was <5; Test type: Other; p < 0.0001, One-sample t-test, 1 sided; The p-value from this test was used to determine the importance of continued treatment in this study. P-value is one-sided with alpha = 0.05

5. Secondary Outcome: Retreatment Efficacy: Change From Time of Retreatment to 12 Weeks After Retreatment in UAS7 Among Participants Randomized to Placebo and Who Were Retreated With Open-Label Omalizumab After Randomization
Description: The UAS is a composite diary-recorded score with numeric severity ratings (0=none to 3=intense) for the number of wheals per 24 hours and the intensity of the pruritus. The total UAS score ranges from 0 to 6. UAS7 is the sum of the daily average UASs (average of morning and evening scores), ranging from 0 to 42 per week. A higher score indicates worse disease. A negative change in score indicates improvement.
Time Frame: At start of retreatment (any time between Weeks 24 and Week 48) and 12 weeks after retreatment (up to Week 60)
Population: Analysis was performed on participants in mITT population who were randomized to placebo arm and who were retreated with open-label omalizumab after randomization. Here, 'Number Analyzed' signifies number of participants with available data for this outcome at specified time-point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (Randomized Participants)
Number analyzed (Participants) | 19
units on a scale
  UAS7 at the Time of Retreatment | 30.51 (8.831)
  Change at 12 Weeks After Retreatment: number analyzed (Participants) | 18
  Change at 12 Weeks After Retreatment | -29.48 (9.632)
Statistical Analysis 1: Comparison: Placebo (Randomized Participants); The null hypothesis for this test was that the mean change from the time of retreatment to 12 weeks after retreatment in UAS7 was zero and the alternative hypothesis was that this change was non-zero; Test type: Other; p < 0.0001, One-sample t-test, 2 sided; The p-value from this test was used to evaluate the importance of retreatment after experiencing clinical worsening

ADVERSE EVENTS:
Time Frame: From start of study drug until 112 days (approximately 5 drug half-lives) after the last dose of study drug or study discontinuation/termination, whichever is later (up to Week 64)
Description: Analysis was performed on safety evaluable population.
Arm/Group | Omalizumab (Non-Randomized Participants) | Omalizumab (Randomized Participants) | Placebo (Randomized Participants)
All-Cause Mortality (participants affected / at risk) | 0/71 | 0/81 | 0/53
Serious Adverse Events (participants affected / at risk) | 0/71 | 2/81 | 3/53
Other Adverse Events (participants affected / at risk) | 22/71 | 28/81 | 22/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Omalizumab (Non-Randomized Participants) (N=71) | Omalizumab (Randomized Participants) (N=81) | Placebo (Randomized Participants) (N=53)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Omalizumab (Non-Randomized Participants) (N=71) | Omalizumab (Randomized Participants) (N=81) | Placebo (Randomized Participants) (N=53)
Fatigue (General disorders) | 0 | 1 | 3
Viral upper respiratory tract infection (Infections and infestations) | 3 | 10 | 6
Upper respiratory tract infection (Infections and infestations) | 2 | 6 | 3
Bronchitis (Infections and infestations) | 1 | 2 | 3
Headache (Nervous system disorders) | 5 | 6 | 3
Urticaria (Skin and subcutaneous tissue disorders) | 10 | 6 | 3
Angioedema (Skin and subcutaneous tissue disorders) | 3 | 4 | 3
Chronic spontaneous urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 3
Prostatomegaly (Reproductive system and breast disorders) | 1/18 | 0/21 | 0/13 — The participants at risk for this sex-specific adverse event were male participants and not all participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2016-05-09): https://cdn.clinicaltrials.gov/large-docs/24/NCT02392624/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-26): https://cdn.clinicaltrials.gov/large-docs/24/NCT02392624/SAP_001.pdf